CLINICAL TRIAL: NCT06692517
Title: Benchmarks in Elective Laparoscopic Cholecystectomy - a National Registry Study
Brief Title: Benchmarks in Elective Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ebba Kihlstedt Pasquier, Principal investigator, Region Östergötland
Other Study IDs: 2022-04311-01
Record Dates: First submitted 2024-05-03; First posted 2024-11-18 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Gall Stone; Gallbladder Inflammation; Gall Bladder Pain; Gallstone; Gall Stones (& [Calculus - Gall Bladder])
Keywords: Laparoscopic cholecystectomy; Benchmarking; Surgical Outcomes; Reference values; Quality Improvement; Risk factors of surgical complications
MeSH Terms: conditions — Gallstones; Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective cholecystectomy: Elective cholecystectomy. Patients with recurrent gallstone attacks, previous cholecystitis, previous cholangitis, or previous pancreatitis. ERCP may be involved if a gallstone is detected in the common bile duct perioperatively.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy

SUMMARY:
The aim of this observational cohort study is to define peri- and postoperative reference values for elective laparoscopic cholecystectomy, using the achievable benchmarks of care methodology (ABC™). Another aim is to develop adjusted reference values for groups with a risk factor of severe postoperative complications. The over-arching aim is to inspire quality improvement initiatives.

DETAILED DESCRIPTION:
The data source is the Swedish patient registry GallRiks, a prospective quality registry for gallbladder surgery and endoscopic retrograde cholangio-pancreatography (ERCP). The time frame will be 2015-2023. Register variables related to surgical quality will be analyzed, such as postoperative complications, perioperative adverse events, surgical duration and length of stay. The study will analyze data for the time of surgery and up to 30 days afterwards. Since the data is not yet available to the researchers the number of enrolled study participants can not be specified with certitude; therefore an anticipated number is given.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years of age
* laparoscopic primary cholecystectomy

Exclusion Criteria:

* patients with current acute cholecystitis, pancreatitis or cholangitis
* cholecystectomy due to malignancy
* other organ surgery performed at the same occasion
* previous upper gastrointestinal surgery
* single port access
* robotic surgery
* no data concerning surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with gall stone disease and, or previous gallbladder inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Benchmark values of elective laparoscopic cholecystectomy | Day of surgery
  The study will use the ABC methodology to identify reference values of surgical duration (minutes), perioperative cholangiography, conversion to open surgery and adverse events
Postoperative benchmark values of elective laparoscopic cholecystectomy | 0-30 days after surgery
  The study will use the ABC methodology to identify reference values of the postoperative variables: hospital length of stay (days), abscess/infection, bleeding, biliary leakage, readmission, reoperation

SECONDARY OUTCOMES:
Adjusted benchmarks for severe complications | 0-30 days after surgery
  Univariable and multivariable logistic regression analysis will be performed to detect any risk factor for severe complications after laparoscopic cholecystectomy. The factors to be investigated are body mass index (kg/m2), age (years), gender, smoking, cardiovascular disease, pulmonary disease, diabetes, immunosuppressive treatment, and treatment with anticoagulants. Adjusted benchmarks will be calculated for factor(s) that in multivariable logistic regression analysis are identified as individual risk factor(s).

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request.